CLINICAL TRIAL: NCT02159807
Title: Randomized Double-blinded Study Designed to Optimize the Dose of Bupivacaine in Combined Spinal Epidurals to Reduce the Incidence of Fetal Bradycardia and Maternal Hypotension
Brief Title: Optimizing Dose of Bupivacaine in Combined Spinal Epidurals To Reduce Side Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 13-0210
Record Dates: First submitted 2014-06-06; First posted 2014-06-10 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Pregnancy
Keywords: Pain control; labor; epidural; pregnant
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1.25 mg Bupivacaine (Active Comparator): 1.25mg of bupivacaine dose with 20 mcg of fentanyl was injected in the spinal portion of the anesthetic
  Interventions: Drug: Bupivacaine; Drug: Fentanyl
- 1.66 mg Bupivacaine (Active Comparator): 1.66mg of bupivacaine dose with 20 mcg of fentanyl was injected in the spinal portion of the anesthetic
  Interventions: Drug: Bupivacaine; Drug: Fentanyl
- 2.5 mg Bupivacaine (Active Comparator): 2.5mg of bupivacaine dose with 20 mcg of fentanyl was injected in the spinal portion of the anesthetic
  Interventions: Drug: Bupivacaine; Drug: Fentanyl

INTERVENTIONS:
Drug: Bupivacaine — The dose of bupivacaine administered intrathecally during placement of the spinal anesthetic.
  Other Names: Fentanyl
Drug: Fentanyl — 20 micrograms routinely administered in combination in the spinal anesthetic

SUMMARY:
The purpose of this study is to determine what dose of medication administered through a combined spinal epidural (CSE) provides the optimal pain relief with the minimal amount of side effects. The 3 doses studied here (1.25, 1.66 and 2.5mg) are routinely use on the labor floor (depending on the physician preference) but the idea is to quantify safety, efficacy and side effects for each of these doses.

DETAILED DESCRIPTION:
A combined spinal epidural (CSE), which is the investigators' customary method of providing pain relief during your labor, is the identification of the epidural space in your lower back with a needle, followed by passing a thinner and longer needle through the first needle. This second needle will enter the patient's "spinal" (intrathecal) space by passing through the dura (thin covering separating the epidural space from the spinal space). The spinal (intrathecal) space is identified by flow of spinal fluid. The dura is the envelope around the spinal cord and the intrathecal space which is filled with spinal fluid. Medication will be injected at once into the spinal space, the thinner needle removed and a fine tube (catheter) will be threaded through the first needle into the epidural space. This catheter is in the epidural space and medication can be given through this catheter later on (hence the term combined) if needed. This study is a comparison of three different dosages (1.25mg, 1.66mg and 2.5 mg) of the local anesthetic (Bupivacaine) that we frequently use in the spinal, mixed with 20 mcg of Fentanyl (also routinely used in standard of care practice), and of its effects on the patient's blood pressure (risk of maternal's drop of the blood pressure with possible bad effects on the blood flow to the baby), on the patient's baby's heart rate (risk of slowing down of the baby heart rate as a consequence of decreased blood flow to the baby), and the patient's pain relief (higher dose of medications are usually more effective for maternal pain relief but have side effects that can be bad for the mother and the baby). The doses of Bupivacaine the investigator routinely use on the labor and delivery floor go from 1.25 to 2.5 mg depending on clinician preferences. These doses are considered standard of care in the literature.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists Physical status) 1-2 parturients at term requesting labor analgesia
* between 37 and 42 weeks gestational age
* maternal age of 18 years or greater

Exclusion Criteria:

* Parturients with pre-eclampsia
* History of pregnancy induced hypertension
* Patients in whom a spinal anesthetic is contraindicated (e.g. coagulopathy, local infection) or those in whom a CSE cannot be performed
* Patients with non reassuring fetal heart rate tracings prior to placement of the CSE

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2015-04-24 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2017-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Epstein, M.D., Principal Investigator — Mount Sinai Roosevelt Hospital
Locations (1):
- Roosevelt hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment period from April 2015 and completed Dec 2017
Groups:
- 1.25 mg Bupivacaine: 1.25mg, mixed with 20 mcg of Fentanyl (also routinely used in standard of care practice), administered intrathecally during placement of the spinal anesthetic. Syringes will be prepared in advance by pharmacy Twenty micrograms of fentanyl is routinely administered in combination with bupivacaine in the spinal
- 1.66 mg Bupivacaine: 1.66mg, mixed with 20 mcg of Fentanyl (also routinely used in standard of care practice), administered intrathecally during placement of the spinal anesthetic. Syringes will be prepared in advance by pharmacy. Twenty micrograms of fentanyl is routinely administered in combination with bupivacaine in the spinal
- 2.5 mg Bupivacaine: 2.5mg, mixed with 20 mcg of Fentanyl (also routinely used in standard of care practice), administered intrathecally during placement of the spinal anesthetic. Syringes will be prepared in advance by pharmacy. Twenty micrograms of fentanyl is routinely administered in combination with bupivacaine in the spinal
Period: Overall Study
Arm/Group | 1.25 mg Bupivacaine | 1.66 mg Bupivacaine | 2.5 mg Bupivacaine
Started | 67 | 52 | 51
Completed | 66 | 51 | 48
Not Completed | 1 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 1
Not completed — No CSF | 1 | 1 | 1
Not completed — elevated blood pressure | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1.25 mg Bupivacaine | 1.66 mg Bupivacaine | 2.5 mg Bupivacaine | Total
Number analyzed (Participants) | 66 | 51 | 48 | 165
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 66 | 51 | 48 | 165
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 51 | 48 | 165
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Fetal Heart Rate (FHR) [Mean (Standard Deviation); unit: beats per min] | 141.13 (12.34) | 136.08 (9.8) | 135.23 (9.57) | 137.48 (10.57)
Pain Score [Mean (Standard Deviation); unit: units on a scale] — Pain Visual Analog Score is from 0-10, with higher score indicating more pain
  units on a scale | 8.15 (2.27) | 8.24 (1.61) | 8.61 (1.51) | 8.33 (1.79)

OUTCOME MEASURES:

1. Primary Outcome: Maternal Blood Pressure
Description: Maternal diastolic blood pressure at 60 minutes after epidural to measure maternal hypotension
Time Frame: at 1 hour
Measure: Mean (Standard Deviation); unit: mm/Hg
Arm/Group | 1.25 mg Bupivacaine | 1.66 mg Bupivacaine | 2.5 mg Bupivacaine
Number analyzed (Participants) | 66 | 51 | 48
mm/Hg | 78.2 (8.17) | 79.58 (9.25) | 80.52 (8.51)

2. Secondary Outcome: Fetal Heart Rate at 1 Hour
Description: Baby's heart rate recorded with the external monitor that is placed on patient's belly, for a duration of 60 minutes after the placement of the combined spinal epidural.
Time Frame: at 1 hour
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | 1.25 mg Bupivacaine | 1.66 mg Bupivacaine | 2.5 mg Bupivacaine
Number analyzed (Participants) | 66 | 51 | 48
beats per minute | 134.73 (10.87) | 137.64 (10.35) | 135.57 (10.07)

3. Secondary Outcome: Mean Change in Visual Analog Scale for Pain
Description: Mean change of her pain relief from the spinal epidural 60 minutes after she received it, using a VAS, scored from 0 to 10, with higher score indicating more pain.
Time Frame: baseline and 60 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.25 mg Bupivacaine | 1.66 mg Bupivacaine | 2.5 mg Bupivacaine
Number analyzed (Participants) | 66 | 51 | 48
score on a scale | 0.43 (1.13) | 0.46 (1.28) | 0.26 (1.07)

ADVERSE EVENTS:
Time Frame: 60 minutes
Arm/Group | 1.25 mg Bupivacaine | 1.66 mg Bupivacaine | 2.5 mg Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/51 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/51 | 0/48
Other Adverse Events (participants affected / at risk) | 0/66 | 0/51 | 1/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1.25 mg Bupivacaine (N=66) | 1.66 mg Bupivacaine (N=51) | 2.5 mg Bupivacaine (N=48)
vasovagal response (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT02159807/Prot_SAP_000.pdf